CLINICAL TRIAL: NCT04100447
Title: An Investigator-Sponsored, Open-Label Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of LB1148 for Subjects Undergoing Elective Bowel Resection
Brief Title: A Study to Evaluate the Safety, Tolerability and Efficacy of LB1148 for Subjects Undergoing Elective Bowel Resection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ronald Hurst, MD, FACS (Other)
Responsible Party: Sponsor-Investigator, Ronald Hurst, MD, FACS, Principal Investigator, Centinela Hospital Medical Center
Organization: Centinela Hospital Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LBS-IST-POI-101
Record Dates: First submitted 2019-08-23; First posted 2019-09-24 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Adhesions; Ileus
Keywords: post-operative; abdominal
MeSH Terms: conditions — Tissue Adhesions; Ileus | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, open label, Phase 1 study to evaluate LB1148 for safety, tolerability, and preliminary efficacy in subjects undergoing elective bowel resection. All subjects will receive LB1148 prior to surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment Arm (Experimental): All subjects will receive 1 dose of study drug (split into 2 administrations), over the 12 hours prior to surgery.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — A total of 700 mL of study drug should be completely consumed orally 2-12 hours prior to surgery as a split dose; 350 mL 6-12 hours prior to surgery and the remaining 350 mL 2-6 hours prior to surgery.
  Other Names: LB1148

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and preliminary efficacy of LB1148 in subjects undergoing elective bowel resection. During abdominal surgery, surgeons handle, manipulate, and often make incisions in the bowel. These actions can create bruising, lesions, and microscopic damage to the bowel, which may allow digestive enzymes to cross the intestinal mucosal barrier potentially resulting in injury both locally and remotely. Leaking digestive enzymes may delay return of normal gastrointestinal (GI) function, lead to a lack of motility in the intestine (ileus), and promote the formation of intestinal scar tissue (adhesions).

DETAILED DESCRIPTION:
The intestinal mucosal barrier plays a key role in both acute critical care medical conditions as well as burdensome chronic diseases. Healthy maintenance of the intestinal mucosal barrier requires oxygenation and blood flow and avoidance of mechanical or physical injury. Potent digestive enzymes are maintained within the intestine as long as normal blood flow continues and no damage or disturbances to the wall occur.

Breakdown of the intestinal mucosal barrier can be produced by wide variety of events. These include prolonged low blood pressure (e.g. during shock), disruption of blood flow (e.g. during ischemia), and physical and mechanical perturbations (e.g. during trauma or abdominal surgery).

One of the key advances toward the use of LB1148 to reduce postoperative complications was the learning that with more subtle perturbations of the mucosal barriers, such as during abdominal surgery, intraluminal pancreatic digestive enzymes played a role in GI dysfunction. Perioperative oral administration of LB1148 in preclinical models was sufficient to reduce the delayed return of GI function. Furthermore, the reduction in pancreatic digestive enzyme-induced tissue damage resulted in a profound reduction in postoperative adhesion formation. Together, these preclinical studies provide evidence that blocking pancreatic digestive enzymes with LB1148 in the intestine reduces local tissue damage, preserves GI function, and reduces adhesion formation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for participation in the study only if they meet ALL of the following inclusion criteria:

  1. Scheduled to undergo an elective (non-emergent) bowel resection. This includes any subject in which a resection of the small intestine, colon, or rectum is performed for any elected indication.
  2. The subject has been informed of the nature of the study, agrees to its provisions, and has provided written informed consent.

Exclusion Criteria:

* Subjects will not be eligible for participation in the study if they meet ANY of the following exclusion criteria:

  1. Subjects who are < 18 or > 85 years of age.
  2. Subjects who require emergency bowel surgery.
  3. Subjects who have had 2 or more abdominal surgeries, excluding the current, for inflammatory bowel disease (IBD), including, but not limited to, IBD, Crohn's Disease, or ulcerative colitis. Note: This does not apply to previous surgeries such as hernia repair unrelated to IBD.
  4. Subjects who meet the American Society of Anesthesiologists (ASA) definition for Class 4 or 5 disease.
  5. Known inability to take the study drug orally (i.e. complete small bowel obstruction).
  6. Subjects with contraindications or potential risk factors to taking TXA. These include:

     1. Known sensitivity to TXA
     2. Recent craniotomy (past 30 days)
     3. Active cerebrovascular bleed
     4. Active thromboembolic disease (such as deep vein thrombosis, pulmonary embolism, cerebral thrombosis, ischemic stroke, or acute coronary syndrome)
     5. Acute promyelocytic leukemia taking all-trans retinoic acid for remission induction
     6. Continuing use of a combined hormonal contraceptive and/or combined hormonal replacement therapy (including combined hormonal pill, patch, or vaginal ring).
  7. Subjects who have the following risk factors for thromboembolic disease:

     1. Known medical history of congenital or acquired thrombophilia such as, but not limited to:

        * Sickle cell disease
        * Nephrotic syndrome
        * Factor V Leiden
        * Prothrombin gene mutation
        * Protein C or S deficiency
        * Antithrombin III deficiency
        * Antiphospholipid syndrome
     2. Neurologic paresis, partial paralysis, or paralysis
     3. Presence of a pacemaker
     4. History of pulmonary embolism, deep vein thrombosis, cerebrovascular accident, or retinal venous/arterial occlusion.
  8. History of or current seizure disorder.
  9. Subjects with myeloproliferative disorders.
  10. Subjects with a Body Mass Index (BMI) > 40.
  11. Any other condition that, in the opinion of the Investigator, would preclude the subject from being an appropriate candidate for the study, including severe renal or hepatic impairment.
  12. Planned treatment with alvimopan (Entereg®) during study participation period.
  13. Subjects who have received any other investigational therapy within 4 weeks.
  14. Subjects with a history of chronic opioid usage, defined by the American Pain Society as daily or near-daily use of opioids for at least 90 days.
  15. Female subjects of childbearing potential with a positive urine or serum pregnancy test or who are not taking (or not willing to take) acceptable birth control measures (abstinence, intrauterine device, contraceptive implant or barrier method) through Study Day 30. Additionally, those women who are lactating and insist on breast feeding within 5 days of the last dose of study drug, are excluded.
  16. Subjects with a known history of radiation enteritis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2020-03-20 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
The number of participants who experience treatment-emergent adverse events (TEAEs) | From first study drug dosing through Day 30
  The number of participants who experience treatment-emergent adverse events (TEAEs) with Investigator-specified relationship to LB1148 and assessment of severity

SECONDARY OUTCOMES:
Number of participants who require a nasogastric (NG) tube placement | During hospitalization (up to 14 days postoperatively), yes or no
  Necessity for nasogastric (NG) tube placement
Average length of time an NG tube was in place, if required | During hospitalization (up to 14 days postoperatively), in hours
  Time NG tube was in place, if needed
Number of participants who experience post surgical vomiting | During hospitalization (from surgical closure to up to 14 days postoperatively), yes or no
  Presence of postsurgical vomiting
Average number of vomiting episodes, when present | During hospitalization (from surgical closure to up to 14 days postoperatively), number of total episodes
  Number of vomiting episode(s)
Average time to first flatus following surgery | During hospitalization (from surgical closure to up to 14 days postoperatively), in hours
  Time to first flatus
Average time to first bowel movement following surgery | During hospitalization (from surgical closure to up to 14 days postoperatively), in hours
  Time to first bowel movement
Average time to tolerate a liquid diet following surgery | During hospitalization (from surgical closure to up to 14 days postoperatively), in hours
  Time to toleration of a liquid diet
Average time to tolerate a solid diet after surgery | During hospitalization (from surgical closure to up to 14 days postoperatively), in hours
  Time to toleration of a solid diet
Average time to hospital discharge order | During hospitalization (from admission to up to 14 days postoperatively), in hours
  Time to hospital discharge order written

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hurst, MD, Principal Investigator — Centinela Hospital Medical Center
Locations (1):
- Centinela Hospital Medical Center, Inglewood, California, United States

IPD SHARING:
Plan to Share IPD: No